CLINICAL TRIAL: NCT01786954
Title: A Comparative Study of Icare Rebound Tonometry With Other Tonometry Modalities in Patients Following Vitreoretinal Surgery.
Brief Title: iCare vs Tonopen vs Goldmann Applanation Post-vitrectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00036498
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-01

CONDITIONS: Intraocular Pressure
Keywords: vitreoretinal surgery; intraocular pressure; applanation; rebound; tonometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Icare then Goldmann then Tonopen (Experimental): Enrolled patients will be subjected to intraocular pressure measurement using Icare rebound tonometry, Tonopen applanation, and Goldmann applanation. Patients receive Icare first and then are randomized to receive Tonopen followed by Goldmann OR Goldmann followed by Tonopen. This arm is Icare then Goldmann then Tonopen.
  Interventions: Device: Icare rebound tonometry; Device: Tonopen applanation; Device: Goldmann applanation
- Icare then Tonopen then Goldmann (Experimental): Enrolled patients will be subjected to intraocular pressure measurement using Icare rebound tonometry, Tonopen applanation, and Goldmann applanation. Patients receive Icare first and then are randomized to receive Tonopen followed by Goldmann OR Goldmann followed by Tonopen. This arm is Icare then Tonopen then Goldmann.
  Interventions: Device: Icare rebound tonometry; Device: Tonopen applanation; Device: Goldmann applanation

INTERVENTIONS:
Device: Icare rebound tonometry
Device: Tonopen applanation
  Other Names: Tonopen Avia
Device: Goldmann applanation

SUMMARY:
The purpose of the study is to compare the measurement of pressure inside the eye using three different FDA-approved devices (Icare, Tonopen, and Goldmann applanation).

DETAILED DESCRIPTION:
The three above devices will be used to measure intraocular pressure in patients one day following vitreoretinal surgery. The underlying reason for surgery is not being considered in this study. The measured pressures will be compared across devices in eyes filled with fluid, gas, and silicone oil.

ELIGIBILITY:
Inclusion Criteria:

* Duke Eye Center patients 18 years or older
* capacity to give legally effective consent
* scheduled to undergo vitreoretinal surgery

Exclusion Criteria:

* individuals unable to give consent
* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hahn, MD, PhD, Principal Investigator — Duke University Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Icare Then Goldmann Then Tonopen: Enrolled patients will be subjected to intraocular pressure measurement using Icare rebound tonometry then Goldmann applanation then Tonopen applanation.
  Icare rebound tonometry
  Goldmann applanation
  Tonopen applanation
- Sequence 2: Icare Then Tonopen Then Goldmann: Enrolled patients will be subjected to intraocular pressure measurement using Icare rebound tonometry then Tonopen applanation then Goldmann applanation.
  Icare rebound tonometry
  Tonopen applanation
  Goldmann applanation
Period: Overall Study
Arm/Group | Sequence 1: Icare Then Goldmann Then Tonopen | Sequence 2: Icare Then Tonopen Then Goldmann
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Icare, Goldmann, Tonopen: Enrolled patients will be subjected to intraocular pressure measurement using Icare rebound tonometry, Tonopen applanation, and Goldmann applanation.
  Icare rebound tonometry
  Tonopen applanation
  Goldmann applanation
Arm/Group | Icare, Goldmann, Tonopen
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Intraocular Pressure
Description: The primary outcome is the measurement of intraocular pressure on postoperative day #1 following vitreoretinal surgery.
Time Frame: postoperative day #1
Population: Of the 68 patients enrolled, only 50 patients who received IOP measurement one day following vitrectomy surgery were analyzed. Those with IOP measurement following non-vitrectomy surgery were subsequently excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Icare: Enrolled patients will be subjected to intraocular pressure measurement using Icare rebound tonometry, Tonopen applanation, and Goldmann applanation.
  Icare rebound tonometry
- Tonopen; Goldmann: Enrolled patients will be subjected to intraocular pressure measurement using Icare rebound tonometry, Tonopen applanation, and Goldmann applanation.
Arm/Group | Icare | Tonopen | Goldmann
Number analyzed (Participants) | 50 | 50 | 50
mm Hg | 15.9 (8.9) | 16.0 (7.3) | 16.9 (7.2)

2. Secondary Outcome: Adverse Events
Description: The secondary outcome is the onset of any adverse events related to measurement of intraocular pressure.
Time Frame: postoperative day #1
Population: Adverse events were analyzed for all enrolled patients, in contrast to IOP measurements, which were only analyzed for the 50 post-vitrectomy patients.
Measure: Number; unit: adverse events
Arm/Group | Icare | Tonopen | Goldmann
Number analyzed (Participants) | 68 | 68 | 68
adverse events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: All patients were examined with a complete ophthalmic exam following IOP measurements.
Groups:
- Sequence 1: Icare, Goldmann, Tonopen: Sequence 1: Icare, then Goldmann, then Tonopen
- Sequence 2: Icare, Tonopen, Goldmann: Sequence 2: Icare, then Tonopen, then Goldmann
Arm/Group | Sequence 1: Icare, Goldmann, Tonopen | Sequence 2: Icare, Tonopen, Goldmann
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No